CLINICAL TRIAL: NCT04541641
Title: Clinical Evaluation of Stability of Implants Placed in Partially Edentulous Maxilla With Poor Bone Quality Via New Reverse Drilling Technique Versus Osteotome Technique: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Stability of Implants Placed in Partially Edentulous Maxilla With Poor Bone Quality Via New Reverse Drilling Technique Versus Osteotome Technique.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mostafa Magdy Awad, doctorate candidate, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PER6-3-1
Record Dates: First submitted 2020-07-27; First posted 2020-09-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Dental Implant

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- osteotome group (Experimental)
  Interventions: Procedure: osteotome technique
- New Reverse Drilling technique (Experimental)
  Interventions: Procedure: New Reverse Drilling technique

INTERVENTIONS:
Procedure: New Reverse Drilling technique — a new technique of dental implant drilling that promote osseodensification by rotating the drills anti-clockwise rather than clockwise to promote bone condensation rather than bone cutting
  Arms: New Reverse Drilling technique
Procedure: osteotome technique — a technique for dental implant placement by using the osteotome to condense the bone and create an osteotome rather than cutting the bone
  Arms: osteotome group

SUMMARY:
The study will compare between osteotome technique and New Reverse Drilling Technique in the placement of dental implant in posterior maxilla , primary outcome will be Implant stability that will be measured by Periotest device . follow up for 6 month.

secondary outcomes will be crestal bone loss , pain and swelling.

ELIGIBILITY:
Inclusion criteria:

1. Partially edentulous patients in the maxillary posterior region.
2. Systemically healthy patient.
3. Presence of proper inter-arch space for placement of the implant prosthetic part.
4. Sufficient bone height and width for implant placement (bone height ≥10mm and bone width ≥6mm).
5. Non-smoker.
6. Patients who are ≥ 20 years old.
7. Good oral hygiene.
8. Acceptance of a one year follow-up period.
9. Informed consent is provided by the patient.

Exclusion criteria:

1. Patients with systemic conditions that may interfere with implant stability,
2. Patients with local pathological defects related to the area of interest.
3. Unmotivated, uncooperative patients with poor oral hygiene.
4. Patients with habits that may jeopardize the implant longevity and affect the results of the study such as alcoholism or parafunctional habits.
5. Inadequate inter-arch space for implant prosthetic part

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2020-10-01 (Estimated); Primary Completion 2022-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
implant stability | 6 months
  the stability of the dental implant when placed in the maxilla of the patient and it will be measured by periotest

SECONDARY OUTCOMES:
crestal bone loss | 6 monthz
  amount of bone loss around the implant . measured in MM with CBVT radiograph

IPD SHARING:
Plan to Share IPD: Undecided